CLINICAL TRIAL: NCT05352113
Title: Intradermal Needle Therapy for Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Collaborators: The Zhejiang Provincial Tongde Hospital (Unknown); The Affiliated Hangzhou First People's Hospital (Unknown)
Responsible Party: Principal Investigator, Xiaomei Shao, Prof, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022ZX010-MDD
Record Dates: First submitted 2022-04-27; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Acupuncture; Randomized controlled clinical trial
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupuncture + SSRIs group (Experimental): This group will include 40 patients with MDD who will be treated with acupuncture and SSRIs antidepressants. Acupoints related to MDD will be stimulated. The oral dose of SSRIs antidepressants will be determined by the clinical specialist.
  Interventions: Drug: SSRIs; Procedure: acupuncture
- acupuncture + placebo group (Experimental): This group will include 40 patients with MDD who will be treated with acupuncture and a placebo. Acupoints related to MDD will be stimulated. The oral dose of SSRIs antidepressants will be determined by the clinical specialist.
  Interventions: Procedure: acupuncture; Drug: placebo
- sham acupuncture + SSRIs group (Experimental): This group will include 40 patients with MDD who will be treated with sham acupuncture and SSRIs antidepressants. The sham acupuncture will be needled on the points 1cm lateral to acupoints. The oral dose of SSRIs antidepressants will be determined by the clinical specialist.
  Interventions: Drug: SSRIs; Procedure: sham acupuncture

INTERVENTIONS:
Drug: SSRIs — SSRIs antidepressants will be used and the oral dose will be determined by the clinical specialist. Once-daily for 6 weeks.
  Other Names: SSRIs antidepressants
  Arms: acupuncture + SSRIs group; sham acupuncture + SSRIs group
Procedure: acupuncture — This study will use the intradermal needle as an acupuncture intervention. Acupoints related to MDD will be stimulated. According to the position of the acupoints, choose a needle of φ0.20*1.5m or φ0.20*1.2mm. Press the needle to insert the acupoint vertically and retain it in the skin. After the intervention, the needle will be retained for 72 hours with a day of rest after removal. During needle retention, participants will be instructed to press the acupoints 3-4 times a day for about 1 minute each time, with the amount of stimulation as much as the patient can tolerate, at an interval of about 4 hours. A total of 10 treatment sessions will be performed for 6 weeks.
  Other Names: intradermal needle
  Arms: acupuncture + SSRIs group; acupuncture + placebo group
Procedure: sham acupuncture — Sham acupuncture will use the same size, color, and material as the verum intradermal needle with a thin silicone pad in the middle instead of the needle body. The sham acupuncture will be needled on the points 1cm lateral to MDD-related acupoints. After the intervention, the needle will be retained for 72 hours with a day of rest after removal. A total of 10 sessions will be performed for 6 weeks.
  Other Names: sham intradermal needle
  Arms: sham acupuncture + SSRIs group
Drug: placebo — Oral placebo mimicking SSRIs antidepressants. Once-daily for 6 weeks.
  Other Names: placebo mimicking SSRIs antidepressants
  Arms: acupuncture + placebo group

SUMMARY:
Major depressive disorder (MDD) is a common mental disorder that affects patients' physical health and quality of life. Although traditional acupuncture therapy has certain advantages in improving MDD, there are still some limitations, such as being time-consuming and some people having a fear of acupuncture. Therefore, intradermal needle therapy will be chosen in the treatment of MDD in this study, which is more convenient, shallow needling, and gentle than traditional acupuncture therapy. The study is designed to investigate the therapeutic effect and safety of intradermal needles for MDD.

DETAILED DESCRIPTION:
A total of 120 participants with MDD who meet the inclusion criteria will be included in the study. Participants will be randomly divided into the SSRIs + acupuncture group, acupuncture + placebo group, and SSRIs + sham acupuncture group. This study will evaluate the efficacy and safety of the intradermal needle for MDD and investigate whether the intradermal needle reduces side effects and increases the efficacy of selective serotonin reuptake inhibitors (SSRIs) antidepressants for MDD. Furthermore, the study will demonstrate whether the intradermal needle has a synergistic effect with SSRIs on the treatment of MDD.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients should meet the diagnostic criteria of the International Classification of Diseases 10th Edition (ICD-10) diagnostic criteria for depression and are evaluated as moderate or severe MDD according to the severity of depression; 2. 12 ≤ age ≤60, male or female; 3. Participants have clear consciousness and could communicate with others normally; 4. Participants could understand the full study protocol and have high adherence. Written informed consent is signed by themselves or their lineal kin (for minor participants, their guardian should sign the informed consent form for them).

Exclusion Criteria:

* 1. Participants with serious primary diseases of cardiovascular, respiratory, digestive, urinary, hematological, endocrine, neurological disease, and other serious primary diseases, and the disease cannot be effectively controlled clinically; 2. Major depressive disorders caused by organic mental disorders, schizophrenia, bipolar disorder, psychoactive substances, and non-addictive substances; 3. Participants with suicidal tendencies; 4. Pregnant or lactating participants; 5. Participants taking other antidepressants that were not SSRIs or the pharmacological effects of such antidepressants have not been cleared; 6. Participants with intellectual disabilities who cannot cooperate with the questionnaire survey; 7. Participants with bleeding tendency, skin disease, allergic constitution, and allergic to adhesive tape; 8. Participants are participating in other trials.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Hamilton Depression Scale-17 (HAMD-17) | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  The HAMD scale is the most commonly used in the clinical assessment of depression, including 17 items. The higher the score, the more severe the depression. 0-7 means no depressive symptoms, 8-17 means mild depression, 18-24 was divided into moderate depression, and 25-52 was divided into severe depression.

SECONDARY OUTCOMES:
Change in the Treatment Emergent SymptomScale (TESS) | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  The TESS scale rated each symptom on three dimensions: severity, the relationship between the symptom and the medication, and the measure taken.
Change in the MOS item short from health survey (SF-36) | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  The SF-36 scale evaluates the quality of healthy life into 8 dimensions, which are divided into two categories: physical health and mental health, namely physical function (PF), role physical (RP), body pain (BP), general health (GH), vitality (VT), social function (SF), role emotional (RE), mental health (MH).
Change in the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  The PSQI is used to assess the sleep quality of the participant in the last 1 month and consisted of 19 self-rated and 5 other rated items. The higher the score, the worse the sleep quality. Sleep quality is divided into 4 levels according to the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei M Shao, Ph.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- Xiaomei Medical Shao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No